CLINICAL TRIAL: NCT01578499
Title: A Randomized, Open-Label, Phase 3 Trial of Brentuximab Vedotin(SGN-35) Versus Physician's Choice (Methotrexate or Bexarotene) in Patients With CD30-Positive Cutaneous T-Cell Lymphoma
Brief Title: A Phase 3 Trial of Brentuximab Vedotin(SGN-35) Versus Physician's Choice (Methotrexate or Bexarotene) in Participants With CD30-Positive Cutaneous T-Cell Lymphoma (ALCANZA Study)
Acronym: ALCANZA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C25001; 2010-024215-14 (EudraCT Number)
Record Dates: First submitted 2012-03-27; First posted 2012-04-17 (Estimated); Results first posted 2018-03-16 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Primary Cutaneous Anaplastic Large Cell Lymphoma; Mycosis Fungoides; Cutaneous T-Cell Lymphoma
Keywords: Brentuximab vedotin; ALCANZA
MeSH Terms: conditions — Lymphoma, Primary Cutaneous Anaplastic Large Cell; Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous | interventions — Brentuximab Vedotin; Methotrexate; Bexarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brentuximab vedotin (Experimental): Brentuximab vedotin 1.8 mg/kg, intravenous over approximately 30 minutes, once on Day 1 of each 21-day cycle and may continue as monotherapy for up to a total of 16 cycles (48 weeks).
  Interventions: Drug: Brentuximab Vedotin
- Methotrexate or Bexarotene (Active Comparator): Methotrexate 5 to 50 mg, tablets, orally, once weekly (dose adjustment is guided by patient response and toxicity) or Bexarotene 300 mg/m^2, tablets, orally, once daily with meals for up to 48 weeks.
  Interventions: Drug: Methotrexate; Drug: Bexarotene

INTERVENTIONS:
Drug: Brentuximab Vedotin — Brentuximab vedotin intravenous injection.
  Other Names: SGN-35
  Arms: Brentuximab vedotin
Drug: Methotrexate — Methotrexate tablets.
  Arms: Methotrexate or Bexarotene
Drug: Bexarotene — Bexarotene tablets.
  Arms: Methotrexate or Bexarotene

SUMMARY:
The purpose of this study is to determine objective response rate (ORR), lasting at least 4 months (ORR4), with brentuximab vedotin in participants with cluster of differentiation antigen 30 positive (CD30+) cutaneous T-cell lymphoma [mycosis fungoides (MF) and primary cutaneous anaplastic large cell lymphoma (pcALCL) ]compared to that achieved with therapy in the control arm.

DETAILED DESCRIPTION:
The drug being tested in this study is called brentuximab vedotin. Brentuximab vedotin is being tested to treat people who have CD30+ cutaneous T-cell lymphoma (mycosis fungoides and primary cutaneous anaplastic large cell lymphoma). This study will look at the overall response of people who took brentuximab vedotin compared to people who took methotrexate or bexarotene as standard care.

The study enrolled 131 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Methotrexate 5 to 50 mg or Bexarotene 300 mg/m^2 (as per physician's choice)
* Brentuximab vedotin 1.8 mg/kg

This multicenter trial is being conducted worldwide. The overall time to participate in this study is approximately 6 years. Participants will make multiple visits to the clinic every 12 weeks for a minimum of 24 months after the end of treatment (EOT) visit, and then every 6 months until death, study closure, or 6 years after enrollment of the last participant.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary consent form
* Male or female participants 18 years or older with diagnosis of mycosis fungoides (MF) or primary cutaneous anaplastic large cell lymphoma (pcALCL)
* Participants with pcALCL who have received prior radiation therapy or at least 1 prior systemic therapy; participants with MF who have received at least 1 prior systemic therapy
* Histologically confirmed CD30+ disease by central laboratory assessment and pathology review
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Female participants who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant
* Male participants who agree to practice effective barrier contraception or agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant
* Clinical laboratory values as specified in protocol
* A 3-week washout period is required from previous treatments (with the exception of a 12-week washout for antibody-directed or immunoglobulin-based immune therapy, or other monoclonal antibody therapies), unless it is not in the best interest of the patient in the opinion of the investigator. Individual cases should be discussed with the project clinician before enrollment.

Exclusion Criteria:

* A concurrent diagnosis of systemic ALCL, or other non Hodgkin lymphoma (excluding LyP) or Sezary syndrome or B2 disease
* Participants with cardiovascular conditions specified in protocols
* Participants with history of another primary malignancy not in remission for at least 3 years
* Known active cerebral/meningeal disease, including signs or symptoms of progressive multifocal leukoencephalopathy (PML);
* Known human immunodeficiency virus (HIV) infection, hepatitis B or Hepatitis C infection
* Oral retinoid therapy for any indication within 3 weeks of study entry
* Corticosteroid therapy within 3 weeks or immunosuppressive chemotherapy or any antibody-directed or immunoglobulin-based immune therapy (e.g., immunoglobulin replacement, other monoclonal antibody therapies) within 12 weeks of first dose of study drug
* Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 of any cycle
* Previous receipt of brentuximab vedotin Please note that there are additional inclusion and exclusion criteria. The study center will determine if you meet all of the criteria.

Site personnel will explain the trial in detail and answer any question you may have if you do qualify for the study. You can then decide whether or not you wish to participate. If you do not qualify for the trial, site personnel will explain the reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-06-11 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2018-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (41):
- United States (8):
  - Los Angeles, California
  - Palo Alto, California
  - Chicago, Illinois
  - Boston, Massachusetts
  - Hackensack, New Jersey
  - New York, New York
  - Pittsburgh, Pennsylvania
  - Houston, Texas
- Australia (5):
  - Concord, New South Wales
  - South Brisbane, Queensland
  - Adelaide, South Australia
  - Nedlands, Western Australia
  - East Melbourne
- Austria (2):
  - Sankt Pölten
  - Vienna
- Leuven, Belgium
- São Paulo, Brazil
- France (5):
  - Nantes
  - Paris
  - Pessac
  - Pierre-Bénite
  - Reims
- Germany (6):
  - Kiel
  - Krefeld
  - Mainz
  - Mannheim
  - Minden
  - Würzburg
- Italy (3):
  - Bologna
  - Florence
  - Meldola
- Warsaw, Poland
- Spain (3):
  - Pamplona, Navarre
  - Barcelona
  - Madrid
- Zurich, Switzerland
- United Kingdom (5):
  - Leeds, West Yorkshire
  - Birmingham
  - Glasgow
  - London
  - Manchester

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Horwitz SM, Scarisbrick JJ, Dummer R, Whittaker S, Duvic M, Kim YH, Quaglino P, Zinzani PL, Bechter O, Eradat H, Pinter-Brown L, Akilov OE, Geskin L, Sanches JA, Ortiz-Romero PL, Weichenthal M, Fisher DC, Walewski J, Trotman J, Taylor K, Dalle S, Stadler R, Lisano J, Bunn V, Little M, Prince HM. Randomized phase 3 ALCANZA study of brentuximab vedotin vs physician's choice in cutaneous T-cell lymphoma: final data. Blood Adv. 2021 Dec 14;5(23):5098-5106. doi: 10.1182/bloodadvances.2021004710. PMID 34507350
- [Derived] Kim YH, Prince HM, Whittaker S, Horwitz SM, Duvic M, Bechter O, Sanches JA, Stadler R, Scarisbrick J, Quaglino P, Zinzani PL, Wolter P, Eradat H, Pinter-Brown LC, Ortiz-Romero PL, Akilov OE, Trotman J, Taylor K, Weichenthal M, Walewski J, Fisher D, McNeeley M, Gru AA, Brown L, Palanca-Wessels MC, Lisano J, Onsum M, Bunn V, Little M, Trepicchio WL, Dummer R. Response to brentuximab vedotin versus physician's choice by CD30 expression and large cell transformation status in patients with mycosis fungoides: An ALCANZA sub-analysis. Eur J Cancer. 2021 May;148:411-421. doi: 10.1016/j.ejca.2021.01.054. Epub 2021 Mar 29. PMID 33794441
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956
- [Derived] Dummer R, Prince HM, Whittaker S, Horwitz SM, Kim YH, Scarisbrick J, Quaglino P, Zinzani PL, Wolter P, Eradat H, Pinter-Brown L, Sanches JA, Ortiz-Romero PL, Akilov OE, Geskin L, Huen A, Walewski J, Wang Y, Lisano J, Richhariya A, Feliciano J, Zhu Y, Bunn V, Little M, Zagadailov E, Dalal MR, Duvic M. Patient-reported quality of life in patients with relapsed/refractory cutaneous T-cell lymphoma: Results from the randomised phase III ALCANZA study. Eur J Cancer. 2020 Jul;133:120-130. doi: 10.1016/j.ejca.2020.04.010. Epub 2020 Jun 2. PMID 32502876
- [Derived] Prince HM, Kim YH, Horwitz SM, Dummer R, Scarisbrick J, Quaglino P, Zinzani PL, Wolter P, Sanches JA, Ortiz-Romero PL, Akilov OE, Geskin L, Trotman J, Taylor K, Dalle S, Weichenthal M, Walewski J, Fisher D, Dreno B, Stadler R, Feldman T, Kuzel TM, Wang Y, Palanca-Wessels MC, Zagadailov E, Trepicchio WL, Zhang W, Lin HM, Liu Y, Huebner D, Little M, Whittaker S, Duvic M; ALCANZA study group. Brentuximab vedotin or physician's choice in CD30-positive cutaneous T-cell lymphoma (ALCANZA): an international, open-label, randomised, phase 3, multicentre trial. Lancet. 2017 Aug 5;390(10094):555-566. doi: 10.1016/S0140-6736(17)31266-7. Epub 2017 Jun 7. PMID 28600132
- See also: Related Info — https://www.alcanzaclinicaltrial.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 34 investigative sites in Australia, Belgium, Brazil, France, Germany, Italy, Poland, Spain, Switzerland, United Kingdom, United States from 11 June 2012 to the Primary Completion data of 06 July 2018.
Pre-assignment Details: Participants with a diagnosis of cluster of differentiation antigen 30 (CD30)-Positive Cutaneous T-Cell Lymphoma were enrolled equally in 1 of 2 arms: brentuximab vedotin 1.8 mg/kg or physician's choice (Methotrexate or Bexarotene).
Period: Overall Study
Arm/Group | Brentuximab Vedotin | Methotrexate or Bexarotene
Started | 66 | 65
Safety Population: Treated | 66 | 62
Intent to Treat Population: CD30+ | 64 | 64
Completed | 32 | 22
Not Completed | 34 | 43
Not completed — Reason not Specified | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 10 | 16
Not completed — Death | 20 | 25
Not completed — Died and End of Study Page not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included participants who received at least 1 dose of study drug, analyzed according to the actual treatment received (n=66,62). Intent-to-treat population (ITT) population included all participants who were identified as CD30+ by the Ventana anti-CD30 (Ber-H2) assay and were randomized to treatment (n=64,64).
Groups:
- Total: Total of all reporting groups
Arm/Group | Brentuximab Vedotin | Methotrexate or Bexarotene | Total
Number analyzed (Participants) | 66 | 64 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Safety population included participants who received at least 1 dose of study drug, analyzed according to the actual treatment received.
  years
    number analyzed (Participants) | 66 | 62 | 128
    (all) | 59.4 (13.80) | 56.6 (14.43) | 58.0 (14.12)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety population included participants who received at least 1 dose of study drug, analyzed according to the actual treatment received.
  Participants
    number analyzed (Participants) | 66 | 62 | 128
    Female | 33 | 28 | 61
    Male | 33 | 34 | 67
Race/Ethnicity, Customized [Number; unit: participants] — Population: ITT population included all participants who were identified as CD30+ by the Ventana anti-CD30 (Ber-H2) assay and were randomized to treatment.
  participants
    White: number analyzed (Participants) | 64 | 64 | 128
    White | 56 | 53 | 109
    Black or African American: number analyzed (Participants) | 64 | 64 | 128
    Black or African American | 3 | 3 | 6
    Asian: number analyzed (Participants) | 64 | 64 | 128
    Asian | 1 | 5 | 6
    Not reported: number analyzed (Participants) | 64 | 64 | 128
    Not reported | 3 | 1 | 4
    Other: number analyzed (Participants) | 64 | 64 | 128
    Other | 1 | 2 | 3
Race/Ethnicity, Customized [Number; unit: participants] — Population: ITT population included all participants who were identified as CD30+ by the Ventana anti-CD30 (Ber-H2) assay and were randomized to treatment.
  participants
    Hispanic or Latino: number analyzed (Participants) | 64 | 64 | 128
    Hispanic or Latino | 2 | 6 | 8
    Not Hispanic or Latino: number analyzed (Participants) | 64 | 64 | 128
    Not Hispanic or Latino | 60 | 50 | 110
    Not reported: number analyzed (Participants) | 64 | 64 | 128
    Not reported | 2 | 8 | 10
Region of Enrollment [Count of Participants; unit: Participants] — Population: Safety population included participants who received at least 1 dose of study drug, analyzed according to the actual treatment received.
  Participants
    Australia: number analyzed (Participants) | 66 | 62 | 128
    Australia | 12 | 8 | 20
    Belgium: number analyzed (Participants) | 66 | 62 | 128
    Belgium | 4 | 2 | 6
    France: number analyzed (Participants) | 66 | 62 | 128
    France | 4 | 3 | 7
    Germany: number analyzed (Participants) | 66 | 62 | 128
    Germany | 3 | 2 | 5
    Italy: number analyzed (Participants) | 66 | 62 | 128
    Italy | 12 | 6 | 18
    Poland: number analyzed (Participants) | 66 | 62 | 128
    Poland | 2 | 1 | 3
    Spain: number analyzed (Participants) | 66 | 62 | 128
    Spain | 2 | 3 | 5
    Switzerland: number analyzed (Participants) | 66 | 62 | 128
    Switzerland | 3 | 3 | 6
    United Kingdom: number analyzed (Participants) | 66 | 62 | 128
    United Kingdom | 8 | 15 | 23
    United States: number analyzed (Participants) | 66 | 62 | 128
    United States | 14 | 17 | 31
    Brazil: number analyzed (Participants) | 66 | 62 | 128
    Brazil | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an Objective Response That Lasts at Least 4 Months (ORR4)
Description: ORR4 was determined by an Independent Review Facility (IRF) based on Global Response Score (GRS) which consisted of a skin assessment by the investigator using the modified severity-weighted assessment tool (mSWAT), nodal and visceral radiographic assessment by an IRF and for the participants with mycosis fungoides (MF) only, detection of circulation Sezary cells. Participants whose first response occurred after the start of subsequent anticancer therapy were excluded. Response Criteria was based on International Society for Cutaneous Lymphomas (ISCL), United States Cutaneous Lymphoma Consortium (USCLC) and Cutaneous Lymphoma Task Force (CLTF) of the European Organisation for Research and Treatment of Cancer (EORTC) Consensus guidelines (Olsen, 2011).
Time Frame: Each Cycle until disease progression, death End of treatment (Median overall follow-up 38.8 months)
Population: The ITT population included all participants who were identified as CD30+ by the Ventana anti-CD30 (Ber-H2) assay and were randomized to treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin | Methotrexate or Bexarotene
Number analyzed (Participants) | 64 | 64
percentage of participants | 54.7 [42.5 to 66.9] | 12.5 [4.4 to 20.6]
Statistical Analysis 1: Comparison: Brentuximab Vedotin vs Methotrexate or Bexarotene; Based on a two-sided Χ² test with a significance level of 0.05, and a 10% dropout rate, a sample size of approximately 124 participants was calculated to provide 90% power to detect a 30% improvement in ORR4 in the brentuximab vedotin group; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value was stratified by baseline disease diagnosis (pcALCL and MF); Risk Difference (RD) = 42.2, 95% CI 2-sided [27.5 to 56.8]

2. Secondary Outcome: Percentage of Participants Achieving a CR
Description: Complete Response (CR) was determined by the IRF based on Global Response Score (GRS) which consisted of a skin assessment by the investigator using the modified severity-weighted assessment tool (mSWAT), nodal and visceral radiographic and for the participants with mycosis fungoides (MF) only, detection of circulation Sezary cells. Response Criteria was based on ISCL, USCLC and CLTF of the EORTC Consensus guidelines (Olsen, 2011).
Time Frame: Each Cycle until disease progression, death or data cutoff (Median overall follow-up 38.8 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin | Methotrexate or Bexarotene
Number analyzed (Participants) | 64 | 64
percentage of participants | 17.2 [7.9 to 26.4] | 1.6 [0.0 to 8.4]
Statistical Analysis 1: Comparison: Brentuximab Vedotin vs Methotrexate or Bexarotene; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel — P-value was stratified by baseline disease diagnosis (pcALCL and MF); Risk Difference (RD) = 15.6, 95% CI 2-sided [-2.5 to 33.0]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was assessed by the IRF and is defined as the time from randomization until disease progression or death due to any cause, whichever occurs first. Disease progression was based on ISCL, USCLC and CLTF of the EORTC Consensus guidelines (Olsen, 2011).
Time Frame: Until disease progression, death or data cutoff (Median PFS follow-up of 38.8 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin | Methotrexate or Bexarotene
Number analyzed (Participants) | 64 | 64
months | 16.7 [15.4 to 21.6] | 3.5 [2.4 to 4.6]
Statistical Analysis 1: Comparison: Brentuximab Vedotin vs Methotrexate or Bexarotene; Test type: Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.378, 95% CI 2-sided [0.247 to 0.577]; Hazard ratio brentuximab vedotin/ comparator (methotrexate or bexarotene) with the 95% CI from a stratified Cox regression model with treatment as the explanatory variable and baseline disease diagnosis (MF or pcALCL) as stratification factor

4. Secondary Outcome: Maximum Change From Baseline in Symptom Domain Score of the Skindex-29 Questionnaire
Description: Skindex-29 is a 29-item dermatology-specific health-related quality of life (HRQoL). The Skindex-29 incorporates a 28-day recall period and consists of 3 domains: symptoms, emotions, and functioning. The domain scores and an overall score are expressed on a 100-point scale, from 0 to 100 with higher scores indicating lower levels of health- HRQoL. A negative change (reduction) from Baseline indicates improvement.
Time Frame: Baseline up to End of Treatment (Week 52)
Population: The ITT population included all participants who were identified as CD30+ by the Ventana anti-CD30 (Ber-H2) assay and were randomized to treatment. Here number of participants analyzed are participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brentuximab Vedotin | Methotrexate or Bexarotene
Number analyzed (Participants) | 58 | 54
score on a scale | -28.08 (26.863) | -8.62 (17.013)
Statistical Analysis 1: Comparison: Brentuximab Vedotin vs Methotrexate or Bexarotene; P-value is calculated using the analysis of covariance (ANCOVA) model controlling for baseline symptom domain score, eastern cooperative oncology group (ECOG) performance status score (=0 and ≥1), and disease diagnosis (pcALCL and MF) between the brentuximab vedotin and comparator (methotrexate or bexarotene) arms; Test type: Superiority or Other; p < 0.001, ANCOVA; Estimate of difference = -19.0, 95% CI 2-sided [-26.7 to -11.4]

5. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was assessed by the IRF in participants with confirmed response [CR or Partial Response (PR)] and is defined as the time between first documentation of response and disease progression. Response Criteria was based on ISCL, USCLC and CLTF of the EORTC Consensus guidelines (Olsen, 2011).
Time Frame: Until disease progression, death or data cutoff (Median follow-up 38.8 months)
Population: The ITT population included all participants who were identified as CD30+ by the Ventana anti-CD30 (Ber-H2) assay and were randomized to treatment. Responders in ITT population were analyzed in this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin | Methotrexate or Bexarotene
Number analyzed (Participants) | 42 | 13
months | 15.1 [9.8 to 25.5] | 18.4 [3.5 to NA] — Upper limit of Confidence Interval (CI) was not estimable due to low number of participants with events.

6. Secondary Outcome: DOR of Skin Response
Description: Duration of skin response (CR and PR) was assessed by the investigator and is defined as the time between the first skin response to progressive disease in skin. Per mSWAT, CR is defined as 100% clearance of skin lesions. PR is defined as 50%-99% clearance of skin disease from Baseline; No new tumors in participants without tumors at Baseline -MF; No new tumors-primary cutaneous anaplastic large cell lymphoma (pcALCL).Progressive disease is defined as ≥ 25% increase in skin disease from baseline, or loss of response: in those with CR or PR, increase of skin score of greater than the sum of nadir plus 50% baseline score, or new tumors in participants without tumors at baseline (MF).
Time Frame: Until disease progression, death or data cutoff (Median follow-up 38.8 months)
Population: The ITT population included all participants who were identified as CD30+ by the Ventana anti-CD30 (Ber-H2) assay and were randomized to treatment. Skin responders in ITT population were analyzed in this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin | Methotrexate or Bexarotene
Number analyzed (Participants) | 47 | 19
months | 18.9 [15.0 to 25.7] | 18.3 [3.5 to NA] — Upper limit of Confidence Interval (CI) was not estimable due to low number of participants with events.

7. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS was assessed by the IRF and is defined as the time from randomization until any cause of treatment failure: disease progression, discontinuation of treatment for any reason, or death due to any cause, whichever occurs first. Disease progression was based on ISCL, USCLC and CLTF of the EORTC Consensus guidelines (Olsen, 2011).
Time Frame: From randomization until disease progression, death or data cutoff (Median follow-up 36.8 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin | Methotrexate or Bexarotene
Number analyzed (Participants) | 64 | 64
months | 9.4 [5.9 to 11.7] | 2.3 [1.7 to 3.5]

8. Secondary Outcome: Cmax: Maximum Observed Concentration for Brentuximab Vedotin
Time Frame: Day 1 pre-dose and 30 minutes after infusion in Cycles 1 and 3
Population: The pharmacokinetic (PK) population included participants with sufficient dose and PK data to reliably estimate PK parameters as determined by a clinical pharmacologist. Here 'Number analyzed' is the number of participants with evaluable data at the specified time-point.
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- pcALCL: Brentuximab Vedotin: Participants with primary cutaneous anaplastic large cell lymphoma (pcALCL) received brentuximab vedotin 1.8 mg/kg, intravenous over approximately 30 minutes, once on Day 1 of each 21-day cycle and may continue as monotherapy for up to a total of 16 cycles (48 weeks).
- MF: Brentuximab Vedotin 1.8 mg/kg: Participants with mycosis fungoides (MF) received brentuximab vedotin 1.8 mg/kg, intravenous over approximately 30 minutes, once on Day 1 of each 21-day cycle and may continue as monotherapy for up to a total of 16 cycles (48 weeks).
Arm/Group | pcALCL: Brentuximab Vedotin | MF: Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 16 | 50
ug/mL
  Cycle 1 Day 1: number analyzed (Participants) | 15 | 50
  Cycle 1 Day 1 | 38.36 (9.427) | 38.40 (8.912)
  Cycle 3 Day 1: number analyzed (Participants) | 12 | 41
  Cycle 3 Day 1 | 40.14 (12.697) | 36.69 (14.249)

9. Secondary Outcome: Ctrough: Observed Concentration at the End of a Dosing Interval for Brentuximab Vedotin
Time Frame: Day 1 pre-dose of Cycles 2 and 4
Population: The PK population included participants with sufficient dose and PK data to reliably estimate PK parameters as determined by a clinical pharmacologist. Here 'Number analyzed' is the number of participants with evaluable data at the specified time-point.
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- pcALCL: Brentuximab Vedotin: Participants with pcALCL received brentuximab vedotin 1.8 mg/kg, intravenous over approximately 30 minutes, once on Day 1 of each 21-day cycle and may continue as monotherapy for up to a total of 16 cycles (48 weeks).
- MF: Brentuximab Vedotin 1.8 mg/kg: Participants with MF received brentuximab vedotin 1.8 mg/kg, intravenous over approximately 30 minutes, once on Day 1 of each 21-day cycle and may continue as monotherapy for up to a total of 16 cycles (48 weeks).
Arm/Group | pcALCL: Brentuximab Vedotin | MF: Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 16 | 50
ug/mL
  Cycle 2 Day 1: number analyzed (Participants) | 11 | 31
  Cycle 2 Day 1 | 3.57 (10.101) | 0.58 (0.517)
  Cycle 4 Day 1: number analyzed (Participants) | 8 | 28
  Cycle 4 Day 1 | 0.99 (0.528) | 0.78 (0.446)

10. Secondary Outcome: Cmax: Maximum Observed Concentration for Monomethyl Auristatin (MMAE) for Brentuximab Vedotin
Time Frame: Day 1 pre-dose and 30 minutes after infusion ended in Cycles 1 and 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | pcALCL: Brentuximab Vedotin | MF: Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 16 | 50
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 13 | 46
  Cycle 1 Day 1 | 2.53 (1.382) | 3.34 (1.901)
  Cycle 3 Day 1: number analyzed (Participants) | 12 | 36
  Cycle 3 Day 1 | 2.96 (1.176) | 3.08 (1.276)

11. Secondary Outcome: Ctrough: Observed Concentration at the End of a Dosing Interval for MMAE for Brentuximab Vedotin
Time Frame: Day 1 pre-dose of Cycles 2 and 4
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | pcALCL: Brentuximab Vedotin | MF: Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 16 | 50
ng/mL
  Cycle 2 Day 1: number analyzed (Participants) | 11 | 33
  Cycle 2 Day 1 | 0.11 (0.095) | 0.09 (0.060)
  Cycle 4 Day 1: number analyzed (Participants) | 10 | 34
  Cycle 4 Day 1 | 0.14 (0.113) | 0.11 (0.091)

12. Secondary Outcome: Number of Participants With Antitherapeutic Antibodies (ATA) to Brentuximab Vedotin
Description: Blood was collected and evaluated for ATA and neutralizing ATA in all participants who received brentuximab vedotin to assess immunogenicity.
Time Frame: Baseline up to End of Treatment (Week 52)
Population: The Safety population included participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | pcALCL: Brentuximab Vedotin | MF: Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 16 | 50
participants
  Immunogenicity-evaluable participants | 14 | 46
  Baseline Negative: ATA negative | 8 | 23
  Baseline Negative: ATA positive | 6 | 19
  Baseline Negative: Transiently Positive | 4 | 9
  Baseline Negative: Persistently Positive | 2 | 10
  Baseline Negative: Neutralizing ATA Positive | 4 | 14
  Baseline Positive: ATA Negative | 0 | 1
  Baseline Positive: ATA Positive | 0 | 3
  Baseline Positive: Transiently Positive | 0 | 3
  Baseline Positive: Persistently Positive | 0 | 0
  Baseline Positive: Neutralizing ATA Positive | 0 | 2

13. Secondary Outcome: Change From Baseline in the Skindex-29 Questionnaire Total Score
Description: Skindex-29 is a 29-item dermatology-specific health-related quality of life (HRQoL). The Skindex-29 incorporates a 28-day recall period and consists of 3 domains: symptoms, emotions, and functioning. The domain scores and an overall score are expressed on a 100-point scale, 0 to 100 with higher scores indicating lower levels of health- HRQoL. A negative change (reduction) from Baseline indicates improvement.
Time Frame: Day 1 of Cycles 1, 2, 4, 6, 8, 10, 12, 14, 16, at End of Treatment (EOT) and during posttreatment long treatment follow-up (LTFU) - (Median follow-up 38.8 months)
Population: The ITT population included all participants who were identified as CD30+ by the Ventana anti-CD30 (Ber-H2) assay and were randomized to treatment. Here 'Number analyzed' is the number of participants with evaluable data at the specified time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brentuximab Vedotin | Methotrexate or Bexarotene
Number analyzed (Participants) | 64 | 64
score on a scale
  Change at Cycle 2: number analyzed (Participants) | 55 | 45
  Change at Cycle 2 | -5.44 (11.055) | -2.49 (11.959)
  Change at Cycle 4: number analyzed (Participants) | 49 | 30
  Change at Cycle 4 | -14.60 (17.488) | -6.71 (9.755)
  Change at Cycle 6: number analyzed (Participants) | 40 | 25
  Change at Cycle 6 | -17.59 (17.770) | -5.40 (9.758)
  Change at Cycle 8: number analyzed (Participants) | 37 | 14
  Change at Cycle 8 | -21.73 (18.882) | -7.28 (16.769)
  Change at Cycle 10: number analyzed (Participants) | 35 | 13
  Change at Cycle 10 | -22.47 (21.722) | -3.71 (21.752)
  Change at Cycle 12: number analyzed (Participants) | 25 | 8
  Change at Cycle 12 | -23.37 (21.555) | -5.22 (17.704)
  Change at Cycle 14: number analyzed (Participants) | 25 | 5
  Change at Cycle 14 | -19.72 (20.980) | -7.49 (22.463)
  Change at Cycle 16: number analyzed (Participants) | 22 | 3
  Change at Cycle 16 | -19.35 (18.911) | 0.75 (10.308)
  Change at End of Treatment: number analyzed (Participants) | 47 | 37
  Change at End of Treatment | -16.26 (23.281) | -0.96 (18.973)
  Change at 3-6 months LTFU: number analyzed (Participants) | 2 | 3
  Change at 3-6 months LTFU | -1.07 (3.704) | -9.48 (21.629)
  Change at 6-9 months LTFU: number analyzed (Participants) | 6 | 11
  Change at 6-9 months LTFU | -8.04 (8.800) | -9.68 (17.789)
  Change at 9-12 months LTFU: number analyzed (Participants) | 7 | 10
  Change at 9-12 months LTFU | -7.94 (15.582) | -4.93 (14.516)
  Change at 12-15 months LTFU: number analyzed (Participants) | 25 | 21
  Change at 12-15 months LTFU | -16.21 (18.438) | -11.16 (18.183)
  Change at 15-18 months LTFU: number analyzed (Participants) | 25 | 18
  Change at 15-18 months LTFU | -19.18 (19.475) | -8.53 (12.768)
  Change at 18-21 months LTFU: number analyzed (Participants) | 22 | 17
  Change at 18-21 months LTFU | -19.27 (20.962) | -5.46 (16.679)
  Change at 21-24 months LTFU: number analyzed (Participants) | 18 | 19
  Change at 21-24 months LTFU | -16.60 (19.875) | -6.86 (14.991)
  Change at 24-27 months LTFU: number analyzed (Participants) | 21 | 16
  Change at 24-27 months LTFU | -17.04 (15.982) | -9.05 (23.990)
  Change at 27-30 months LTFU: number analyzed (Participants) | 20 | 18
  Change at 27-30 months LTFU | -12.45 (19.639) | -7.97 (16.401)
  Change at >30 months LTFU: number analyzed (Participants) | 23 | 20
  Change at >30 months LTFU | -11.49 (22.470) | -1.07 (18.886)

14. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy General Questionnaire (FACT-G) Score
Description: FACT-G is a 27-item general cancer QOL instrument completed by participants receiving cancer treatment. FACT-G incorporates a 7-day recall period and contains 4 primary subscales: Physical Well-Being (PWB; sum of 7 items, point range 0-28); Social/Family Well-Being (SWB, sum of 7-items, point range 0-28); Emotional Well-Being (EWB; sum of 6-items, point range 0-24); Functional Well-Being (FWB; sum of 7-items, point range 0-28); Fact-G total score=sum of PWB, SWB, EWB, FWB, point range 0-108. Higher scores for the total scales and subscales indicate better quality of life. A negative change (reduction) from Baseline indicates improvement.
Time Frame: Day 1 of Cycles 1, 2, 4, 6, 8, 10, 12, 14, 16, at EOT and during posttreatment (LTFU) - (Median follow-up 38.8 months)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brentuximab Vedotin | Methotrexate or Bexarotene
Number analyzed (Participants) | 64 | 64
score on a scale
  Change at Cycle 2: number analyzed (Participants) | 56 | 46
  Change at Cycle 2 | 1.43 (10.168) | -0.37 (11.723)
  Change at Cycle 4: number analyzed (Participants) | 50 | 32
  Change at Cycle 4 | 1.75 (12.014) | 1.78 (10.740)
  Change at Cycle 6: number analyzed (Participants) | 40 | 25
  Change at Cycle 6 | 4.23 (14.257) | 2.24 (13.108)
  Change at Cycle 8: number analyzed (Participants) | 37 | 13
  Change at Cycle 8 | 5.96 (16.030) | 2.54 (10.809)
  Change at Cycle 10: number analyzed (Participants) | 35 | 13
  Change at Cycle 10 | 6.61 (16.971) | 4.38 (15.040)
  Change at Cycle 12: number analyzed (Participants) | 27 | 8
  Change at Cycle 12 | 7.94 (18.837) | 8.61 (21.024)
  Change at Cycle 14: number analyzed (Participants) | 26 | 6
  Change at Cycle 14 | 9.04 (14.104) | 10.75 (13.615)
  Change at Cycle 16: number analyzed (Participants) | 22 | 4
  Change at Cycle 16 | 5.08 (9.230) | 7.88 (23.432)
  Change at End of Treatment: number analyzed (Participants) | 47 | 37
  Change at End of Treatment | 0.35 (16.067) | -2.29 (17.171)
  Change at 3-6 months LTFU: number analyzed (Participants) | 2 | 2
  Change at 3-6 months LTFU | 16.00 (18.385) | -2.92 (8.367)
  Change at 6-9 months LTFU: number analyzed (Participants) | 6 | 12
  Change at 6-9 months LTFU | -0.19 (19.648) | -2.59 (12.473)
  Change at 9-12 months LTFU: number analyzed (Participants) | 7 | 10
  Change at 9-12 months LTFU | 3.62 (17.651) | -5.32 (10.555)
  Change at 12-15 months LTFU: number analyzed (Participants) | 26 | 19
  Change at 12-15 months LTFU | 8.33 (14.918) | -1.34 (11.905)
  Change at 15-18 months LTFU: number analyzed (Participants) | 24 | 18
  Change at 15-18 months LTFU | 3.03 (12.618) | 2.94 (14.756)
  Change at 18-21 months LTFU: number analyzed (Participants) | 24 | 16
  Change at 18-21 months LTFU | 3.35 (11.117) | -0.19 (14.316)
  Change at 21-24 months LTFU: number analyzed (Participants) | 17 | 18
  Change at 21-24 months LTFU | 1.51 (5.471) | 0.61 (14.505)
  Change at 24-27 months LTFU: number analyzed (Participants) | 20 | 15
  Change at 24-27 months LTFU | 4.20 (7.952) | 1.42 (17.870)
  Change at 27-30 months LTFU: number analyzed (Participants) | 19 | 17
  Change at 27-30 months LTFU | -1.57 (17.488) | 1.93 (8.716)
  Change at >30 months LTFU: number analyzed (Participants) | 22 | 19
  Change at >30 months LTFU | -6.22 (15.222) | -2.85 (5.518)

15. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AEs and SAEs were assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A SAE is any AE that results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event.
Time Frame: First dose of study drug through 30 days after last dose of study drug (Up to 450 days)
Population: The Safety population included participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Brentuximab Vedotin | Methotrexate or Bexarotene
Number analyzed (Participants) | 66 | 62
participants
  AEs | 63 | 56
  SAEs | 18 | 18

ADVERSE EVENTS:
Time Frame: All-Cause mortality: Baseline up to End of study (Up to 6 years); Serious and Other adverse events: First dose of study drug through 30 days after last dose of study drug (Up to 450 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Brentuximab Vedotin | Methotrexate or Bexarotene
All-Cause Mortality (participants affected / at risk) | 22/66 | 25/62
Serious Adverse Events (participants affected / at risk) | 18/66 | 18/62
Other Adverse Events (participants affected / at risk) | 60/66 | 51/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin (N=66) | Methotrexate or Bexarotene (N=62)
Cellulitis (Infections and infestations) | 2 | 0
Superinfection bacterial (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 3 — One treatment-emergent death occurred in participant with sepsis during treatment with brentuximab vedotin and is not related.
Urosepsis (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 0 | 1
Periorbital infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 2 | 4
Extravasation (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 — One treatment-emergent death occurred in participant with pcALCL during treatment with brentuximab vedotin and is related.
Fatigue (General disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — One treatment-emergent death occurred in participant with lymphoma during treatment with brentuximab vedotin and is not related.
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Stress (Psychiatric disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — One treatment-emergent death occurred in participant with pulmonary embolism during treatment with brentuximab vedotin and is not related.
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin (N=66) | Methotrexate or Bexarotene (N=62)
Peripheral sensory neuropathy (Nervous system disorders) | 31 | 1
Peripheral motor neuropathy (Nervous system disorders) | 4 | 0
Paraesthesia (Nervous system disorders) | 6 | 1
Dysgeusia (Nervous system disorders) | 5 | 0
Headache (Nervous system disorders) | 5 | 6
Dizziness (Nervous system disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 24 | 9
Vomiting (Gastrointestinal disorders) | 11 | 3
Diarrhoea (Gastrointestinal disorders) | 18 | 4
Constipation (Gastrointestinal disorders) | 3 | 5
Fatigue (General disorders) | 18 | 18
Asthenia (General disorders) | 7 | 5
Pyrexia (General disorders) | 9 | 8
Oedema peripheral (General disorders) | 7 | 6
Chills (General disorders) | 4 | 2
Peripheral swelling (General disorders) | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Skin infection (Infections and infestations) | 2 | 6
Urinary tract infection (Infections and infestations) | 4 | 4
Staphylococcal skin infection (Infections and infestations) | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 10 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 11
Weight decreased (Investigations) | 6 | 2
Alanine aminotransferase increased (Investigations) | 3 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 4
Blood cholesterol increased (Investigations) | 0 | 4
Blood triglycerides increased (Investigations) | 0 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 5 | 4
Anaemia (Blood and lymphatic system disorders) | 3 | 6
Hypertension (Vascular disorders) | 6 | 0
Dry eye (Eye disorders) | 0 | 4
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Insomnia (Psychiatric disorders) | 2 | 6
Anxiety (Psychiatric disorders) | 0 | 4
Hypothyroidism (Endocrine disorders) | 0 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 8
Pruritus generalised (Skin and subcutaneous tissue disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT01578499/SAP_000.pdf
  • Study Protocol (2014-12-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT01578499/Prot_001.pdf